CLINICAL TRIAL: NCT00513422
Title: The Effect of Glucosamine Sulphate on Structural Disease Progression in Knee Osteoarthritis and the Cost-effectiveness of Glucosamine Sulphate for Knee Arthritis.
Brief Title: The Long-term Evaluation of Glucosamine Sulphate Study
Acronym: LEGS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sydney (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Dr Marlene Fransen, University of Sydney
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GI-IM-LEGS-L; NHMRC 402511 (Other Grant/Funding Number: National Health and Medical Research Council of Australia); NHMRC 402781 (Other Grant/Funding Number: National Health and Medical Research Council of Australia)
Record Dates: First submitted 2007-08-07; First posted 2007-08-08 (Estimated); Last update posted 2010-06-30 (Estimated); Status verified 2010-06

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis, knee; Glucosamine; Chondroitin; Disease progression; NSAIDs
MeSH Terms: conditions — Osteoarthritis, Knee; Disease Progression | interventions — Glucosamine; Chondroitin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Glucosamine sulfate 1500mg and chondroitin sulfate 800mg (low molecular weight, bovine)
  Interventions: Dietary Supplement: Glucosamine sulphate and chondroitin
- 2 (Experimental): Glucosamine sulfate 1500mg
  Interventions: Dietary Supplement: Glucosamine sulphate
- 3 (Experimental): Chondroitin sulfate 800mg
  Interventions: Dietary Supplement: Chondroitin sulphate
- 4 (Placebo Comparator): Matching glucosamine/chondroitin placebo capsules
  Interventions: Dietary Supplement: Placebo capsules for glucosamine and chondroitin

INTERVENTIONS:
Dietary Supplement: Glucosamine sulphate and chondroitin — Glucosamine: Two 750mg capsules once daily for two years;
  Chondroitin: Two 400mg capsules once daily for two years.
  Other Names: Glucosamine; Chondroitin
  Arms: 1
Dietary Supplement: Glucosamine sulphate — Glucosamine: Two 750mg capsules once daily for two years;
  Placebo Chondroitin: Two capsules once daily for two years.
  Other Names: Glucosamine
  Arms: 2
Dietary Supplement: Chondroitin sulphate — Chondroitin sulphate: Two 400mg capsules once daily for two years;
  Placebo glucosamine: Two capsules once daily for two years.
  Other Names: Chondroitin
  Arms: 3
Dietary Supplement: Placebo capsules for glucosamine and chondroitin — Two placebo glucosamine capsules once daily for two years;
  Two placebo chondroitin capsules once daily for two years.
  Other Names: Double placebo
  Arms: 4

SUMMARY:
The primary aim of this study is to determine if the dietary supplements, glucosamine sulphate and/or chondroitin can limit or reduce structural disease progression whilst providing symptomatic benefit in people with osteoarthritis (OA) of the knee.

The specific hypotheses to be tested in the proposed double blind, placebo-controlled, randomised clinical trial are that, compared to participants allocated to placebo, participants allocated to either or both of these dietary supplements will demonstrate:

* reduced medial tibio-femoral joint space narrowing at 2 years AND;
* reduced knee pain over 1 year

These benefits will be achieved by participants allocated to glucosamine sulphate and/or chondroitin (the study treatments) without concomitant:

* increased use of analgesics
* reduced health-related quality of life
* reduced participation in leisure-time physical activity

DETAILED DESCRIPTION:
The LEGS study is a double blind, placebo-controlled randomised clinical trial using a 2 x 2 factorial design. Participant will be randomly allocated to one of the four possible treatment combinations:

* Glucosamine and Chondroitin (double active)
* Placebo Glucosamine and Chondroitin
* Glucosamine and Placebo Chondroitin
* Placebo Glucosamine and Placebo Chondroitin (double placebo)

Each allocation involves taking 4 study treatment capsules once a day for two years.

A total of 600 participants with symptomatic knee OA will be recruited by general media advertising and by General Practitioners through the New South Wales Divisions of general practice.

ELIGIBILITY:
Inclusion Criteria:

* Knee pain, or taking NSAIDs/ analgesia for knee pain on most days past month
* Knee pain 4-10 on 10cm VAS
* Medial tibio-femoral compartment joint space narrowing in symptomatic knee

Exclusion Criteria:

* Unstable diabetes
* <2mm medial tibio-femoral compartment joint space width

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2007-10; Primary Completion 2011-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Medial tibio-femoral joint space narrowing (mm) | MRI (1 year) Radiographs (2 years)
Knee pain (11 point Likert scale) | Bimonthly for 1 year

SECONDARY OUTCOMES:
WOMAC | 1 year, 2 years
Patients global assessment | Bimonthly for 1 year
Total NSAIDs use | Bimonthly for 1 year
General health status (SF-12v2) | 1 year, 2 years
Cost-effectiveness (cost per OMERACT-OARSI responder) | 2 years
Leisure time physical activity | 1 year, 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Fransen, PhD, MPH, Principal Investigator — University of Sydney, Faculty of Health Sciences; Richard Day, MB, BS, MD, Principal Investigator — University of New South Wales; Charles Bridges-Webb, MB, BS, Principal Investigator — Royal College of General Practitioners; John Edmonds, MB,BS, Principal Investigator — University of New South Wales; Robyn Norton, PhD, MPH, Principal Investigator — The George Institute, University of Sydney; Mark Woodward, PhD, MSc, Principal Investigator — The George Institute, University of Sydney; Lynette March, PhD, MB, BS, Principal Investigator — University of Sydney; Philip Sambrook, MB, BS, Principal Investigator — Institute of Bone and Joint Research, University of Sydney
Locations (1):
- Marlene Fransen, Sydney, New South Wales, Australia

REFERENCES:
- [Derived] Simic M, Harmer AR, Agaliotis M, Nairn L, Bridgett L, March L, Votrubec M, Edmonds J, Woodward M, Day R, Fransen M. Clinical risk factors associated with radiographic osteoarthritis progression among people with knee pain: a longitudinal study. Arthritis Res Ther. 2021 Jun 4;23(1):160. doi: 10.1186/s13075-021-02540-9. PMID 34088340
- [Derived] Fransen M, Agaliotis M, Nairn L, Votrubec M, Bridgett L, Su S, Jan S, March L, Edmonds J, Norton R, Woodward M, Day R; LEGS study collaborative group. Glucosamine and chondroitin for knee osteoarthritis: a double-blind randomised placebo-controlled clinical trial evaluating single and combination regimens. Ann Rheum Dis. 2015 May;74(5):851-8. doi: 10.1136/annrheumdis-2013-203954. Epub 2014 Jan 6. PMID 24395557
- [Derived] Laba TL, Brien JA, Fransen M, Jan S. Patient preferences for adherence to treatment for osteoarthritis: the MEdication Decisions in Osteoarthritis Study (MEDOS). BMC Musculoskelet Disord. 2013 May 6;14:160. doi: 10.1186/1471-2474-14-160. PMID 23647688